CLINICAL TRIAL: NCT07093892
Title: Cohort Study on Cognitive Decline in Elderly
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20250361
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease，Mild Cognitive Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Alzheimer's Disease (AD) prevention and control currently face severe challenges, with limited treatment options and effectiveness available. Once the disease progresses to the AD stage, it is essentially irreversible. Before the onset of AD, there is a prolonged asymptomatic period and a stage of mild cognitive impairment (MCI), which represents a critical window for early screening, diagnosis, and intervention. Therefore, early screening, diagnosis, and intervention during the MCI stage are crucial for slowing or halting the rising trend of AD and alleviating its disease burden.

This study plans to enroll elderly individuals from communities around Peking University Third Hospital to establish a prospective cohort. Participants will undergo cognitive assessments and blood biomarker testing, followed by a three-year follow-up and management program. The study aims to obtain epidemiological data on MCI and AD in community populations, investigate the relationships between known risk factors, genetic factors, and blood biomarkers with disease progression, explore additional biomarkers, and develop predictive models. These efforts will contribute to promoting early diagnosis, early intervention, and improved prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55 years or older;
2. No diagnosis of Alzheimer's disease (AD);
3. Participants are able to complete cognitive tests, provide biological samples, undergo neuroimaging examinations, and cooperate throughout the entire study process;
4. Signed informed consent.

Exclusion Criteria:

1. Participants with severe mental illness, tumor-related cachexia, severe hepatic or renal insufficiency, or other major physical conditions that may hinder cooperation with the examinations;
2. Participants who are unable to complete the required assessments due to visual or hearing impairments;
3. Contraindications for MRI or other study-related examinations.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll elderly individuals meeting the inclusion/exclusion criteria from communities surrounding Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The change of MMSE | 3 years
  MMSE is a 30-point questionnaire used to measure cognitive function
The change of MoCA | 3 years
  MoCA is a 30-point questionnaire used to measure cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Yang, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No